CLINICAL TRIAL: NCT07273461
Title: Investigation of the Effects of Pain Neuroscience Education on Knowledge and Attitudes Toward Pain in Physiotherapy Students
Brief Title: Pain Neuroscience Education in Physiotherapy Students: Effects on Knowledge and Attitudes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ayşe ŞİMŞEK (Other)
Responsible Party: Sponsor-Investigator, Ayşe ŞİMŞEK, Research Assistant, PhD student, Hacettepe University
Organization: Hacettepe University (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: KBU-2025-2154
Record Dates: First submitted 2025-11-27; First posted 2025-12-09 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-11

CONDITIONS: Pain Knowledge; Pain Management; Physiotherapist Students
Keywords: pain neuroscience education; physiotherapy students; pain knowledge; pain beliefs
MeSH Terms: conditions — Agnosia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Pain Neuroscience Education Group (Experimental): Experimental: Pain Neuroscience Education Group Arm Description: Single-group intervention arm receiving a 70-minute Pain Neuroscience Education session. Outcome measures were collected at baseline and immediately after the intervention.
  Interventions: Behavioral: Pain Neuroscience Education (PNE)

INTERVENTIONS:
Behavioral: Pain Neuroscience Education (PNE) — The program consists of a single 70-minute Pain Neuroscience Education (PNE) session, which includes explanations of pain neurophysiology, central sensitization, biopsychosocial pain concepts, and cognitive-behavioral factors influencing chronic pain. Delivered by a trained certified physiotherapist.

SUMMARY:
This study aims to examine the immediate effects of a single-session Pain Neuroscience Education (PNE) program on pain-related knowledge and attitudes among undergraduate physiotherapy students. The PNE session focuses on explaining pain neurophysiology, chronic pain mechanisms, central sensitization, and the biopsychosocial factors that influence pain. Participants complete validated questionnaires assessing pain knowledge, pain-related beliefs, and attitudes before and immediately after the intervention. The purpose of the study is to determine whether a brief educational session can produce immediate improvements in pain knowledge and pain-related attitudes across different academic years in physiotherapy students.

DETAILED DESCRIPTION:
This study is a retrospective registration of a completed pre-post interventional study conducted among undergraduate physiotherapy students. The objective of the research was to evaluate the immediate effects of a single-session Pain Neuroscience Education (PNE) program on pain-related knowledge, beliefs, and attitudes.

The PNE session lasted approximately 70 minutes and was delivered by a physiotherapist trained in pain neuroscience and the biopsychosocial model. The session covered pain neurophysiology, the distinction between acute and chronic pain, central sensitization, factors contributing to pain experiences, and the role of cognition, emotions, and behaviors within the biopsychosocial framework.

Participants completed self-report outcome measures at two time points:

Baseline (pre-intervention)

Immediately after the intervention

Outcome measures included validated instruments assessing pain knowledge and pain-related beliefs:

Revised Neurophysiology of Pain Questionnaire (rNPQ)

Pain Knowledge and Attitudes Questionnaire (KNAP)

Health Care Providers' Pain and Impairment Relationship Scale (HC-PAIRS)

Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT)

The study followed a single-group design with no control group and no randomization.

The study was conducted between April and October 2025 at Karabük University, Turkey. Ethical approval was obtained from the Karabük University Non-Interventional Clinical Research Ethics Committee (Decision No: 2025/2154), and written informed consent was obtained from all participants prior to data collection.

The results of this research aim to contribute to the understanding of how a brief PNE session may provide immediate improvements in pain-related knowledge and attitudes among physiotherapy students. The findings may support the integration of structured pain education approaches into physiotherapy curricula and early clinical training programs.

ELIGIBILITY:
Inclusion Criteria:

* Undergraduate physiotherapy and rehabilitation students (1st, 2nd, 3rd, or 4th year)
* Willing to participate and able to provide written informed consent

Exclusion Criteria:

* Having previously received formal Pain Neuroscience Education (PNE)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 155 (Actual)
Dates: Start 2025-04-01 (Actual); Primary Completion 2025-10-31 (Actual); Study Completion 2025-10-31 (Actual)

PRIMARY OUTCOMES:
Revised Neurophysiology of Pain Questionnaire (rNPQ) | Baseline and immediately after the intervention
  The rNPQ assessed participants' knowledge of pain neurophysiology. The scale measures participants' knowledge level on topics such as pain mechanisms, neuropathic pain, central sensitization, and biopsychosocial components of pain. The scale consists of a total of 12 questions with "true", "false", or "I don't know" answers. Incorrect answers and answers marked as undecided receive 0 points. The scale is scored between 0 and 12, and pain knowledge increases as the score increases.
Knowledge and Attitudes of Pain Questionnaire (KNAP) | Baseline and immediately after the intervention
  Participants' knowledge and attitudes towards pain were measured with the KNAP. The KNAP scale consists of 30 questions and is scored on a six-point Likert scale ranging from completely disagree to completely agree. The total score is between 0 and 150 points. A higher score from the scale indicates knowledge and attitudes that better reflect modern pain neuroscience.
Pain Attitudes and Beliefs Scale for Physiotherapists (PABS-PT) | Baseline and immediately after the intervention
  The PABS-PT was used to distinguish between biomedical and biopsychosocial orientations towards treating low back pain in physiotherapists. The scale is scored as 1 = strongly disagree and 6 = strongly agree. Treatment orientation is measured in biomedical (factor 1) and biopsychosocial (factor 2) subscales. Subscale scores are calculated by simply summing the scores corresponding to the selected response for each item. The subscale with the highest score indicates the participant's dominant treatment orientation
Health Care Providers' Pain Impairment Relationship Scale (HC-PAIRS ) | Baseline and immediately after the intervention
  The HC-PAIRS was developed to examine the impact of attitudes and beliefs of health professionals on the clinical management of chronic nonspecific low back pain.The scale consists of 12 items, ranging from 1 (completely disagree) to 7 (completely agree). After items 1 and 5 are reversed, the total score is calculated and ranges from 12 to 84. Higher scores indicate a strong belief that low back pain is a legitimate cause of activity limitation and disability, and negative attitudes and beliefs of health professionals towards low back pain.

CONTACTS AND LOCATIONS:
Overall Officials: Ayşe Şimşek, MSc, Study Director — Karabuk University
Locations (1):
- Karabük University Faculty of Health Sciences, Karabük, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No